CLINICAL TRIAL: NCT02519335
Title: Use of the Cardioprotectant Dexrazoxane During Congenital Heart Surgery: Proposal for Pilot Investigation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI no longer at this facility
Sponsor: Medical City Children's Hospital (Other)
Collaborators: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCCH-001
Record Dates: First submitted 2015-05-14; First posted 2015-08-10 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2017-03

CONDITIONS: Heart Defects, Congenital
Keywords: cardiopulmonary bypass; ischemia reperfusion injury
MeSH Terms: conditions — Heart Defects, Congenital; Reperfusion Injury | interventions — Dexrazoxane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dexrazoxane (Other): Trial subjects will be assigned preoperatively to receive Dexrazoxane at one of three doses: low (200mg/m2/dose), medium (300mg/m2/dose), or high (400mg/m2/dose). Four patients will be assigned to each dosing regimen for a total of 12 patients.
  The medication will be administered in the operating room 15-30 minutes prior to starting cardiopulmonary bypass (dose #1), after finishing cardiopulmonary bypass (dose #2), and on the morning after surgery in the cardiac intensive care unit (dose #3).
  Interventions: Drug: Dexrazoxane

INTERVENTIONS:
Drug: Dexrazoxane — Dose escalation every 4 subjects from 200mg/m2/dose; 300mg/m2/dose to 400mg/m2/dose
  Other Names: Zinecard

SUMMARY:
Cardiopulmonary bypass and arrest of the heart during cardiac surgery are necessary to allow the surgeon to perform heart operations. However, these processes can cause injury to the heart which may worsen post-operative outcomes. In fact, the effects of these injuries may continue after surgery, and lead to a long-term decrease in heart function. Neonates and young infants are at particular risk for this occurrence.

While much research has been done in adults looking for medicines that might protect the heart during surgery, few studies have been conducted in neonates and young infants. The investigators are testing Dexrazoxane, which has proven to be cardio-protective in pediatric cancer patients, in the hope that it may lessen cardiac injury during and after congenital heart surgery, and thereby improve outcomes in the neonatal and young infant population.

In order to accomplish this, the investigators must first determine how Dexrazoxane can be safely administered to young children with congenital heart disease. Therefore, the investigators are performing a pilot study of 12 children to assess:

1. how Dexrazoxane at 3 different doses is metabolized in the body of a child age 0-6 months during and after congenital heart surgery, and
2. the safety of Dexrazoxane use in the neonatal and young infant population undergoing cardiac surgery.

DETAILED DESCRIPTION:
Neonates and infants undergoing heart surgery with cardioplegic arrest experience both inflammation and myocardial ischemia-reperfusion [IR] injury. These processes provoke myocardial apoptosis and oxygen free radical formation which result in cardiac injury and dysfunction. Dexrazoxane is a derivative of EDTA that is approved for prevention of anthracycline-related cardiotoxicity. It provides cardioprotection through reduction of toxic reactive oxygen species [ROS], and suppression of apoptosis.

The deleterious effects of cardiopulmonary bypass [CPB] with cardioplegic arrest of the heart during congenital heart operations greatly influence postoperative morbidity and mortality. Neonates and infants undergoing cardiac surgery experience both a systemic inflammatory response, and myocardial IR injury as cardioplegic arrest is reversed. These processes provoke elaboration of cytokines and activation of the complement cascade, as well as oxygen free radical formation and induction of myocardial apoptosis (1, 2, 3). Frequently, myocardial injury and cardiac dysfunction ensue, leading to low cardiac output syndrome and multi-system organ failure. The irreversible component of these injuries, in addition to the abnormal workloads imposed on the myocardium from the anatomic defects themselves, may have consequences for long-term cardiac function, and may in part explain contractile dysfunction observed late after congenital heart

The investigators propose a pilot pharmacokinetic/safety trial of dexrazoxane in children 0-6 months of age, followed by a randomized, double-blind, clinical trial of dexrazoxane vs placebo during congenital heart surgery. The investigators will evaluate postoperative time to resolution of organ failure, development of low cardiac output syndrome, length of cardiac ICU and hospital stays, and echocardiographic indices of cardiac dysfunction. Results could establish the safety and clinical utility of dexrazoxane in ameliorating ischemia-reperfusion injury during congenital heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* age 6 months and under
* open heart surgery requiring CPB and use of cardioplegia
* parent/guardian consent for study obtained surgery planned Monday to Friday

Exclusion Criteria:

* gestational age <36weeks
* known syndrome or genetic abnormality, except Trisomy 21 single ventricle physiology
* concurrent enrollment in another research protocol
* no parental/guardian consent obtained
* ECMO utilization prior to surgery or necessary at the time of ICU admission

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Resolution of organ failure | 60 days postoperative
  measured by number of days to the point of being off invasive mechanical ventilation, renal replacement therapy and inotropic support

SECONDARY OUTCOMES:
Postoperative low cardiac output syndrome | 60 days
  observance of clinical signs or symptoms such as tachycardia, oliguria, poor perfusion and cardiac arrest.

OTHER OUTCOMES:
Myocardial injury | 60 days
  determined by elevated serum cardiac troponin
Oxidative stress | 60 days
  measured by lipoperoxidation (serum F2 isoprostane), plasma thiobarbituric acid reactive substance (TBARS), and plasma total antioxidant activity
Inflammatory activation (IL-6 and IL-10) | 60 days
Myocardial dysfunction (via echocardiogram) | 60 days
  measured by Tei index, tissue doppler E/E ratio, and ventricular ejection fraction
Neurologic injury (activin A) | 60 days
  measured by serum activin A concentration
ICU and hospital length of stay | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Stromberg, MD, Principal Investigator — Medical City Children's Hospital
Locations (1):
- Medical City Children's Hospital, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaney MA. Corticosteroids and cardiopulmonary bypass : a review of clinical investigations. Chest. 2002 Mar;121(3):921-31. doi: 10.1378/chest.121.3.921. PMID 11888978
- [Background] Caputo M, Mokhtari A, Rogers CA, Panayiotou N, Chen Q, Ghorbel MT, Angelini GD, Parry AJ. The effects of normoxic versus hyperoxic cardiopulmonary bypass on oxidative stress and inflammatory response in cyanotic pediatric patients undergoing open cardiac surgery: a randomized controlled trial. J Thorac Cardiovasc Surg. 2009 Jul;138(1):206-14. doi: 10.1016/j.jtcvs.2008.12.028. Epub 2009 Feb 23. PMID 19577081
- [Background] Hare JM. Oxidative stress and apoptosis in heart failure progression. Circ Res. 2001 Aug 3;89(3):198-200. No abstract available. PMID 11485969
- [Background] Pasquali SK, Hall M, Li JS, Peterson ED, Jaggers J, Lodge AJ, Marino BS, Goodman DM, Shah SS. Corticosteroids and outcome in children undergoing congenital heart surgery: analysis of the Pediatric Health Information Systems database. Circulation. 2010 Nov 23;122(21):2123-30. doi: 10.1161/CIRCULATIONAHA.110.948737. Epub 2010 Nov 8. PMID 21060075
- [Background] Graham EM, Atz AM, Butts RJ, Baker NL, Zyblewski SC, Deardorff RL, DeSantis SM, Reeves ST, Bradley SM, Spinale FG. Standardized preoperative corticosteroid treatment in neonates undergoing cardiac surgery: results from a randomized trial. J Thorac Cardiovasc Surg. 2011 Dec;142(6):1523-9. doi: 10.1016/j.jtcvs.2011.04.019. Epub 2011 May 20. PMID 21600592
- [Background] Schroeder VA, Pearl JM, Schwartz SM, Shanley TP, Manning PB, Nelson DP. Combined steroid treatment for congenital heart surgery improves oxygen delivery and reduces postbypass inflammatory mediator expression. Circulation. 2003 Jun 10;107(22):2823-8. doi: 10.1161/01.CIR.0000070955.55636.25. Epub 2003 May 19. PMID 12756159
- [Background] Checchia PA, Backer CL, Bronicki RA, Baden HP, Crawford SE, Green TP, Mavroudis C. Dexamethasone reduces postoperative troponin levels in children undergoing cardiopulmonary bypass. Crit Care Med. 2003 Jun;31(6):1742-5. doi: 10.1097/01.CCM.0000063443.32874.60. PMID 12794414
- [Background] Clarizia NA, Manlhiot C, Schwartz SM, Sivarajan VB, Maratta R, Holtby HM, Gruenwald CE, Caldarone CA, Van Arsdell GS, McCrindle BW. Improved outcomes associated with intraoperative steroid use in high-risk pediatric cardiac surgery. Ann Thorac Surg. 2011 Apr;91(4):1222-7. doi: 10.1016/j.athoracsur.2010.11.005. PMID 21440149
- [Background] Clancy RR, McGaurn SA, Goin JE, Hirtz DG, Norwood WI, Gaynor JW, Jacobs ML, Wernovsky G, Mahle WT, Murphy JD, Nicolson SC, Steven JM, Spray TL. Allopurinol neurocardiac protection trial in infants undergoing heart surgery using deep hypothermic circulatory arrest. Pediatrics. 2001 Jul;108(1):61-70. doi: 10.1542/peds.108.1.61. PMID 11433055
- [Background] Jin Z, Duan W, Chen M, Yu S, Zhang H, Feng G, Xiong L, Yi D. The myocardial protective effects of adenosine pretreatment in children undergoing cardiac surgery: a randomized controlled clinical trial. Eur J Cardiothorac Surg. 2011 May;39(5):e90-6. doi: 10.1016/j.ejcts.2010.12.052. Epub 2011 Feb 20. PMID 21342773
- [Background] Ferreira R, Burgos M, Milei J, Llesuy S, Molteni L, Hourquebie H, Boveris A. Effect of supplementing cardioplegic solution with deferoxamine on reperfused human myocardium. J Thorac Cardiovasc Surg. 1990 Nov;100(5):708-14. PMID 2232833
- [Background] Menasche P, Pasquier C, Bellucci S, Lorente P, Jaillon P, Piwnica A. Deferoxamine reduces neutrophil-mediated free radical production during cardiopulmonary bypass in man. J Thorac Cardiovasc Surg. 1988 Oct;96(4):582-9. PMID 2845199
- [Background] Menasche P, Antebi H, Alcindor LG, Teiger E, Perez G, Giudicelli Y, Nordmann R, Piwnica A. Iron chelation by deferoxamine inhibits lipid peroxidation during cardiopulmonary bypass in humans. Circulation. 1990 Nov;82(5 Suppl):IV390-6. PMID 2225430
- [Background] Zheng H, Dimayuga C, Hudaihed A, Katz SD. Effect of dexrazoxane on homocysteine-induced endothelial dysfunction in normal subjects. Arterioscler Thromb Vasc Biol. 2002 Jul 1;22(7):E15-8. doi: 10.1161/01.atv.0000023187.25914.5b. PMID 12117747
- [Background] Junjing Z, Yan Z, Baolu Z. Scavenging effects of dexrazoxane on free radicals. J Clin Biochem Nutr. 2010 Nov;47(3):238-45. doi: 10.3164/jcbn.10-64. Epub 2010 Oct 29. PMID 21103033
- [Background] Popelova O, Sterba M, Haskova P, Simunek T, Hroch M, Guncova I, Nachtigal P, Adamcova M, Gersl V, Mazurova Y. Dexrazoxane-afforded protection against chronic anthracycline cardiotoxicity in vivo: effective rescue of cardiomyocytes from apoptotic cell death. Br J Cancer. 2009 Sep 1;101(5):792-802. doi: 10.1038/sj.bjc.6605192. Epub 2009 Jul 21. PMID 19623174
- [Background] Zhou L, Sung RY, Li K, Pong NH, Xiang P, Shen J, Ng PC, Chen Y. Cardioprotective effect of dexrazoxane in a rat model of myocardial infarction: anti-apoptosis and promoting angiogenesis. Int J Cardiol. 2011 Oct 20;152(2):196-201. doi: 10.1016/j.ijcard.2010.07.015. Epub 2010 Aug 6. PMID 20692056
- [Background] Spagnuolo RD, Recalcati S, Tacchini L, Cairo G. Role of hypoxia-inducible factors in the dexrazoxane-mediated protection of cardiomyocytes from doxorubicin-induced toxicity. Br J Pharmacol. 2011 May;163(2):299-312. doi: 10.1111/j.1476-5381.2011.01208.x. PMID 21232037 (Retraction: PMID 32512636 Br J Pharmacol. 2020 Jul;177(13):3123)
- [Background] Hasinoff BB, Schroeder PE, Patel D. The metabolites of the cardioprotective drug dexrazoxane do not protect myocytes from doxorubicin-induced cytotoxicity. Mol Pharmacol. 2003 Sep;64(3):670-8. doi: 10.1124/mol.64.3.670. PMID 12920203
- [Background] Wiseman LR, Spencer CM. Dexrazoxane. A review of its use as a cardioprotective agent in patients receiving anthracycline-based chemotherapy. Drugs. 1998 Sep;56(3):385-403. doi: 10.2165/00003495-199856030-00009. PMID 9777314
- [Background] Brier ME, Gaylor SK, McGovren JP, Glue P, Fang A, Aronoff GR. Pharmacokinetics of dexrazoxane in subjects with impaired kidney function. J Clin Pharmacol. 2011 May;51(5):731-8. doi: 10.1177/0091270010369675. Epub 2010 May 19. PMID 20484616
- [Background] Lipshultz SE, Rifai N, Dalton VM, Levy DE, Silverman LB, Lipsitz SR, Colan SD, Asselin BL, Barr RD, Clavell LA, Hurwitz CA, Moghrabi A, Samson Y, Schorin MA, Gelber RD, Sallan SE. The effect of dexrazoxane on myocardial injury in doxorubicin-treated children with acute lymphoblastic leukemia. N Engl J Med. 2004 Jul 8;351(2):145-53. doi: 10.1056/NEJMoa035153. PMID 15247354
- [Background] Elbl L, Hrstkova H, Tomaskova I, Michalek J. Late anthracycline cardiotoxicity protection by dexrazoxane (ICRF-187) in pediatric patients: echocardiographic follow-up. Support Care Cancer. 2006 Feb;14(2):128-36. doi: 10.1007/s00520-005-0858-8. Epub 2005 Jul 21. PMID 16034614
- [Background] Sanchez-Medina J, Gonzalez-Ramella O, Gallegos-Castorena S. The effect of dexrazoxane for clinical and subclinical cardiotoxicity in children with acute myeloid leukemia. J Pediatr Hematol Oncol. 2010 May;32(4):294-7. doi: 10.1097/MPH.0b013e3181d321b3. PMID 20404753
- [Background] Choi HS, Park ES, Kang HJ, Shin HY, Noh CI, Yun YS, Ahn HS, Choi JY. Dexrazoxane for preventing anthracycline cardiotoxicity in children with solid tumors. J Korean Med Sci. 2010 Sep;25(9):1336-42. doi: 10.3346/jkms.2010.25.9.1336. Epub 2010 Aug 12. PMID 20808678
- [Background] Tebbi CK, London WB, Friedman D, Villaluna D, De Alarcon PA, Constine LS, Mendenhall NP, Sposto R, Chauvenet A, Schwartz CL. Dexrazoxane-associated risk for acute myeloid leukemia/myelodysplastic syndrome and other secondary malignancies in pediatric Hodgkin's disease. J Clin Oncol. 2007 Feb 10;25(5):493-500. doi: 10.1200/JCO.2005.02.3879. PMID 17290056
- [Background] Barry EV, Vrooman LM, Dahlberg SE, Neuberg DS, Asselin BL, Athale UH, Clavell LA, Larsen EC, Moghrabi A, Samson Y, Schorin MA, Cohen HJ, Lipshultz SE, Sallan SE, Silverman LB. Absence of secondary malignant neoplasms in children with high-risk acute lymphoblastic leukemia treated with dexrazoxane. J Clin Oncol. 2008 Mar 1;26(7):1106-11. doi: 10.1200/JCO.2007.12.2481. PMID 18309945
- [Background] Lipshultz SE, Scully RE, Lipsitz SR, Sallan SE, Silverman LB, Miller TL, Barry EV, Asselin BL, Athale U, Clavell LA, Larsen E, Moghrabi A, Samson Y, Michon B, Schorin MA, Cohen HJ, Neuberg DS, Orav EJ, Colan SD. Assessment of dexrazoxane as a cardioprotectant in doxorubicin-treated children with high-risk acute lymphoblastic leukaemia: long-term follow-up of a prospective, randomised, multicentre trial. Lancet Oncol. 2010 Oct;11(10):950-61. doi: 10.1016/S1470-2045(10)70204-7. Epub 2010 Sep 16. PMID 20850381
- [Background] Vrooman LM, Neuberg DS, Stevenson KE, Asselin BL, Athale UH, Clavell L, Cole PD, Kelly KM, Larsen EC, Laverdiere C, Michon B, Schorin M, Schwartz CL, Cohen HJ, Lipshultz SE, Silverman LB, Sallan SE. The low incidence of secondary acute myelogenous leukaemia in children and adolescents treated with dexrazoxane for acute lymphoblastic leukaemia: a report from the Dana-Farber Cancer Institute ALL Consortium. Eur J Cancer. 2011 Jun;47(9):1373-9. doi: 10.1016/j.ejca.2011.03.022. Epub 2011 Apr 20. PMID 21514146
- [Background] Hoffman TM, Wernovsky G, Atz AM, Kulik TJ, Nelson DP, Chang AC, Bailey JM, Akbary A, Kocsis JF, Kaczmarek R, Spray TL, Wessel DL. Efficacy and safety of milrinone in preventing low cardiac output syndrome in infants and children after corrective surgery for congenital heart disease. Circulation. 2003 Feb 25;107(7):996-1002. doi: 10.1161/01.cir.0000051365.81920.28. PMID 12600913
- [Background] Su XW, Undar A. Brain protection during pediatric cardiopulmonary bypass. Artif Organs. 2010 Apr;34(4):E91-102. doi: 10.1111/j.1525-1594.2009.00963.x. PMID 20420605
- [Background] Vidrio H, Carrasco OF, Rodriguez R. Antivasoconstrictor effect of the neuroprotective agent dexrazoxane in rat aorta. Life Sci. 2006 Dec 14;80(2):98-104. doi: 10.1016/j.lfs.2006.08.025. Epub 2006 Aug 25. PMID 17007888
- [Background] Florio P, Abella RF, de la Torre T, Giamberti A, Luisi S, Butera G, Cazzaniga A, Frigiola A, Petraglia F, Gazzolo D. Perioperative activin A concentrations as a predictive marker of neurologic abnormalities in children after open heart surgery. Clin Chem. 2007 May;53(5):982-5. doi: 10.1373/clinchem.2006.077149. Epub 2007 Mar 15. PMID 17363421
- [Background] Fiser DH. Assessing the outcome of pediatric intensive care. J Pediatr. 1992 Jul;121(1):68-74. doi: 10.1016/s0022-3476(05)82544-2. PMID 1625096
- [Background] Holcenberg JS, Tutsch KD, Earhart RH, Ungerleider RS, Kamen BA, Pratt CB, Gribble TJ, Glaubiger DL. Phase I study of ICRF-187 in pediatric cancer patients and comparison of its pharmacokinetics in children and adults. Cancer Treat Rep. 1986 Jun;70(6):703-9. PMID 3089595
- [Background] Mou SS, Giroir BP, Molitor-Kirsch EA, Leonard SR, Nikaidoh H, Nizzi F, Town DA, Roy LC, Scott W, Stromberg D. Fresh whole blood versus reconstituted blood for pump priming in heart surgery in infants. N Engl J Med. 2004 Oct 14;351(16):1635-44. doi: 10.1056/NEJMoa041065. PMID 15483282